CLINICAL TRIAL: NCT02671032
Title: Characterisation of Audiological Outcomes With the Nucleus CI532 Cochlear Implant in Adult Subjects.
Brief Title: CHANGE Feasibility Study
Acronym: CLTD5626
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: The Hearing Cooperative Research Centre (Other); Royal Victoria Eye and Ear Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTD5626
Record Dates: First submitted 2016-01-27; First posted 2016-02-02 (Estimated); Results first posted 2020-11-20 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Hearing Loss
Keywords: Cochlear Prosthesis Implantation
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implantation with Nucleus CI532 cochlear implant (Experimental): All participants will receive the same treatment - Implantation with Nucleus CI532 cochlear implant.
  Interventions: Device: Nucleus CI532 cochlear implant

INTERVENTIONS:
Device: Nucleus CI532 cochlear implant

SUMMARY:
The purpose of the feasibility study is to examine audiological outcomes (audiometry and speech perception) and safety (adverse events and adverse device effects) with the Nucleus CI532 cochlear implant in group of adult subjects (n=12) who meet current criteria for cochlear implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Meet current cochlear implant indications at the implanting centre
2. In addition to meeting current cochlear implant indications, subjects must also possess preoperative unaided hearing thresholds between 40 to 65 dB HL at 250 & 500Hz in the ear to be implanted.
3. Fluent speaker in the local language used to assess clinical performance
4. Eighteen years of age or older at the time of implantation with no upper age limit

Exclusion Criteria:

1. Evidence of hearing loss prior to 5 years of age.
2. Sensorineural severe-to-profound hearing loss greater than 20 years at 2 kHz and above.
3. Simultaneous bilateral cochlear implantation or prior cochlear implantation in the ear to be implanted.
4. Additional disabilities that may affect the subject's participation or safety during the clinical investigation.
5. Medical or psychological conditions that contraindicate undergoing general anaesthesia or surgery.
6. Ossification, malformation or any other cochlear anomaly, such as common cavity, that might prevent complete insertion of the electrode array, as confirmed by medical examination.
7. Hearing impairment due to lesion or neuropathy of the acoustic nerve, VIII nerve or central auditory pathway.
8. Active middle-ear infection,
9. Tympanic membrane perforation
10. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure(s) and prosthetic devices
11. Unwillingness or inability of the candidate to comply with all investigational requirements.
12. Patients with existing CSF shunts or drains, existing perilymph fistula, skull fracture or CSF leak.
13. Patients with recurrent episodes of bacterial meningitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cowan, DipAud PhD, Principal Investigator — HEARing CRC
Locations (2):
- Australia (2):
  - The Hearing Cooperative Research Centre, Carlton, Victoria
  - Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for sharing IPD. Data may be provided to individual researchers on request.

RESULTS

PARTICIPANT FLOW:
Groups:
- Implantation With Nucleus CI532 Cochlear Implant: All participants will receive the same treatment - Implantation with Nucleus CI532 cochlear implant.
  Nucleus CI532 cochlear implant
Period: Overall Study
Arm/Group | Implantation With Nucleus CI532 Cochlear Implant
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Implantation With Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 63 [23 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 12
Average Initial Age of Hearing Aid Fitted [Mean (Full Range); unit: years] | 45 [12 to 59]
Onset of Initial Hearing Loss [Mean (Full Range); unit: years] | 37 [12 to 48]
Severe Hearing Loss [Count of Participants; unit: Participants] — Severe hearing loss is classified as hearing loss of 66-90 dB
  Participants | 3

OUTCOME MEASURES:

1. Primary Outcome: Report on Degree of Hearing as Measured by Pure Tone Audiogram
Description: unaided audiogram at time intervals indicated above in ear to be implanted and implanted ear.
Time Frame: 6 months and 12 months post activation
Measure: Number; unit: participants
Arm/Group | Implantation With Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 12
participants
  6 months, 250 Hz : Function <= 70 dB HL | 5
  6 months, 250 Hz : Preserved 70 > dB HL <= 90 | 2
  6 months, 250 Hz : Preserved > 90 dB HL | 2
  6 months, 500 Hz : Function <= 70 dB HL | 0
  6 months, 500 Hz : Preserved 70 > dB HL <= 90 | 4
  6 months, 500 Hz : Preserved > 90 dB HL | 4
  6months, 750 Hz : Function <= 70 dB HL | 0
  6months, 750 Hz : Preserved 70 > dB HL <= 90 | 4
  6months, 750 Hz : Preserved > 90 dB HL | 2
  12 months - 250 Hz : Function <= 70 dB HL | 4
  12 months - 250 Hz : Preserved 70 > dB HL <= 90 | 3
  12 months - 250 Hz : Preserved > 90 dB HL | 2
  12 months - 500 Hz : Function <= 70 dB HL | 0
  12 months - 500 Hz : Preserved 70 > dB HL <= 90 | 5
  12 months - 500 Hz : Preserved > 90 dB HL | 3
  12 months - 750 Hz : Function <= 70 dB HL | 0
  12 months - 750 Hz : Preserved 70 > dB HL <= 90 | 4
  12 months - 750 Hz : Preserved > 90 dB HL | 2

2. Primary Outcome: Report on Clinical Performance in Quiet and Noise
Description: Speech perception assessment with monosyllabic words and sentences percentage correct in competing noise at a fixed signal-to-noise ratio (+5dB).
Time Frame: 3 months, 6 months and 12 months post activation
Measure: Mean (Standard Deviation); unit: percentage of correct words
Arm/Group | Implantation With Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 12
percentage of correct words
  Quiet baseline, untreated ear | 22 (15.4)
  Baseline quiet, treated ear | 10.4 (8.7)
  Quiet, electronic alone 3 months | 29.9 (7.9)
  Quiet, electronic alone 6 months | 31.9 (8.7)
  Quiet, electronic alone 12 months | 32.8 (7.8)
  Quiet, hybrid hearing 3 months | 27.4 (9.7)
  Quiet, hybrid hearing 6 months | 27.0 (11.6)
  Quiet, hybrid hearing 12 months | 25.3 (8.1)
  Noise baseline, untreated ear | 48.2 (36.8)
  Noise baseline, treated ear | 25.2 (28.3)
  Noise, electric alone 3 months | 81.7 (17.2)
  Noise, electric alone 6 months | 80.8 (23.2)
  Noise, electric alone 12 months | 85.1 (14.8)
  Noise, hydrid hearing 3 months | 77.5 (18.8)
  Noise, hybrid hearing 6 months | 72.0 (29.3)
  Noise, hybrid hearing 12 months | 83.7 (10.8)

3. Primary Outcome: Report of Medical/Surgical and Device Related Adverse Events.
Description: Report of medical/surgical and device related adverse events compared to current approved labeling with regard to type, frequency and seriousness.
Time Frame: 12 months post activation.
Measure: Number; unit: Adverse Events
Arm/Group | Implantation With Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 12
Adverse Events
  Possibly procedure related - pinna/behind pain | 1
  Possibly procedure related - dizziness | 2
  Possibly procedure related - drop in hearing | 1
  Possibly procedure related - nausea | 1
  Possibly procedure related - right ear tinnitus | 1
  Procedure related - headache | 1
  Procedure related - incision site pain | 1
  Procedure related - incision site tenderness | 1
  Procedure related - jaw ache | 1
  Procedure related - initial insertion tip foldover | 1
  Possibly device related - pinna/behind pain | 1
  Possibly device related - dizziness | 2
  Possibly device related - drop in hearing | 1
  Possibly device related - nausea | 1
  Device related - initial insertion top foldover | 1

4. Secondary Outcome: Report on Patient Reported Outcome Measures for Speech, Spatial and Qualities of Hearing Scale (SSQ)
Description: Effect of intervention (implantation with CI532 cochlear implant) will be assessed by the change in SSQ scores from preoperative to 6 months post activation, where scores follow a system of 0 = not at all and 10 = perfectly in response to questions.
Time Frame: Preoperative and 6 months post activation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implantation With Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 12
score on a scale
  Baseline - Speech Hearing | 4.2 (2.3)
  Baseline - Spatial Hearing | 3.9 (2.1)
  Baseline - Qualities of Hearing | 4.7 (2.3)
  Baseline - Overall SSQ | 4.3 (2.1)
  6 Month - Speech Hearing | 5.9 (2.6)
  6 Month - Spatial Hearing | 5.4 (2.7)
  6 Month - Qualities of Hearing | 6.5 (2.4)
  6 Month - Overall SSQ | 6.0 (2.4)

5. Secondary Outcome: Glasgow Benefit Inventory (GBI).
Description: Effect of intervention (implantation with CI532 cochlear implant) will be assessed at 6 months post activation with the Glasgow Benefit Inventory (GBI). Glasgow Benefit Inventory (GBI) is a measure of patient reported benefit developed especially for otorhinolaryngological interventions where scores range from -100 to 100, where a higher score corresponds to a better benefit outcome and a negative score value corresponds to a worse outcome.
Time Frame: 6 months post activation
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Implantation With Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 12
score on a scale
  General Benefit | 66.7 [0 to 100]
  Social Benefit | 43.1 [0 to 100]
  Physical Benefit | 15.3 [0 to 100]
  Average Benefit | 54 [0 to 100]

ADVERSE EVENTS:
Time Frame: 12 months and 30 days
Arm/Group | Implantation With Nucleus CI532 Cochlear Implant
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 7/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implantation With Nucleus CI532 Cochlear Implant (N=12)
Discomfort/Pain of Pinna and Behind (Ear and labyrinth disorders) | 2 (2)
Onset of tinnitus in right ear (Injury, poisoning and procedural complications) | 1 (1) — Possibly related to procedure
Dizziness (Injury, poisoning and procedural complications) | 3 (3) — Two events possibly related to procedure and/or device
Drop in hearing (Injury, poisoning and procedural complications) | 1 (1) — Possibly related to procedure and/or device
Nausea (Injury, poisoning and procedural complications) | 1 (1) — Possibly related to procedure and/or device
Cold-like symptoms including sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Injury, poisoning and procedural complications) | 2 (2) — One event possibly related to procedure
Jaw ache (Injury, poisoning and procedural complications) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1)
Incision site tenderness (Injury, poisoning and procedural complications) | 1 (1)
Otitis Externa (Ear and labyrinth disorders) | 1 (1)
Vomiting (Nervous system disorders) | 1 (1)
Abscess in left breast (Infections and infestations) | 1 (1)
Polymyalgia Rheumatica (Immune system disorders) | 1 (1)
Arm infection (Infections and infestations) | 1 (1)
Cactus injury to wrist (Injury, poisoning and procedural complications) | 1 (1) — Not related to procedure
Hip pain left and right sides (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in body joints (Musculoskeletal and connective tissue disorders) | 1 (1)
Sun spot removal (actinic keratosis) (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/32/NCT02671032/Prot_SAP_000.pdf